CLINICAL TRIAL: NCT03429530
Title: Study of microRNAs as a Diagnostic Tool for HCV-related Hepatocellular Carcinoma
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: HMHamed (Other)
Responsible Party: Sponsor-Investigator, HMHamed, DR Hager, Assiut University
Organization: Assiut University (Other)
Other Study IDs: miRNA in HCC
Record Dates: First submitted 2018-02-06; First posted 2018-02-12 (Actual); Last update posted 2018-02-12 (Actual); Status verified 2018-02

CONDITIONS: miRna in HCC

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Group1: 20 patients with chronic HCV
- GroupII: 20 patient with chronic HCV related liver cirrhosis
- GroupIII: 40 patients with chronic HCV related liver cirrhosis complicated by hepatocellular cacinoma
- group IV: 20 healthy blood donors will also be included as a control group

SUMMARY:
The aim of this work is to study the role of circulating miRNAs in diagnosis of HCV related hepatocellular carcinoma.

DETAILED DESCRIPTION:
Early diagnosis of hepatocellular carcinoma can significantly improve the overall survival of HCC patients, currently available diagnostic markers are still inadequate and limited by their low sensitivity and specificity. For instance, the gold standard marker, alpha-fetoprotein (AFP), has a false negative rate up to 40% for early stage of HCC. It is worthy to mention that the level of AFP was reported in a normal range of 25% of patients with advanced HCC. These discrepancies suggest the need of discovering new reliable diagnostic markers for patients with HCC. miRNAs are small endogenous, non-coding, ssRNA that are 21-30 nucleotides in length. As for the relationship between miRNA and HCC several studies have demonstrated that the aberrant expression of specific miRNA can be detected in HCC cells and tissues.

miRNAs expression profile analysis has allowed the characterization of 'identity' associated with each type of human cancer and this 'identity' is correlated with carcinogenesis, tumor progression, and response to tumor treatment.

ELIGIBILITY:
Inclusion Criteria:

* RNA extraction and quantitative Real-Time PCR analysis
* Diagnosis of HCV will be based on detection of anti-HCV antibodies
* Diagnosis of liver cirrhosis will be based on ultrasonography, biochemically and elastography when available
* Diagnosis of HCC will be based on ultrasonography, the typical criteria in triphasic multislice CT scan

Exclusion Criteria:

* HBV or autoimmune or metabolic liver disease
* serological evidence of human immunodeficiency virus (HIV) infection
* malignancy in other organs
* After intervention in treatment of hepatocellular carcinoma

Ages: 20 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This study will be carried out in Al-Raghy hospital (Assiut university), in collaboration with Medical Microbiology &Immunology Department.
  Eighty patients with HCV related chronic liver disease will be included. GroupI; 20 patients with chronic HCV GroupII; 20 patient with chronic HCV related liver cirrhosis GroupIII; 40 patients with chronic HCV related liver cirrhosis complicated by hepatocellular cacinoma Control group: (group IV) Sex and age matched 20 healthy blood donors will also be included as a control group
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-02-15 (Estimated); Primary Completion 2019-02 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
the role of circulating miRNAs in diagnosis of HCV related hepatocellular carcinoma. | basline
  cilculating miRNAs in serum samples of HCV related HCC, HCV related liver cirrhosis , chronic HCV and healthy control group